CLINICAL TRIAL: NCT02713217
Title: Adapting and Implementing the Blended Collaborative Care Model in CBOCs
Brief Title: Implementing a Blended Care Model That Integrates Mental Healthcare and Primary Care Using Telemedicine and Care Management for Patients With Depression or Alcohol Use Disorder in Small Primary Care Clinics
Acronym: Tele-PCMHI
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CRE 12-310
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Depressive Disorders; Alcohol Use Disorders; Post-traumatic Stress Disorder (PTSD)
Keywords: depressive disorder; alcohol-related disorders; telemedicine; rural health; collaborative care; post-traumatic stress disorder (PTSD)
MeSH Terms: conditions — Depressive Disorder; Alcoholism; Stress Disorders, Post-Traumatic; Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-Implementation Cohort: Eligible patients will be recruited and enrolled prior to implementation of the blended integrated care model in each study site. They will be exposed to care as usual in the CBOCs.
  Interventions: Other: Usual Care
- Post-Implementation Cohort: Eligible patients will be recruited and enrolled following implementation of the blended integrated care model in each study site. These participants are thus exposed to the "intervention" model.
  Interventions: Other: Blended Telemedicine-Based Integrated Care

INTERVENTIONS:
Other: Usual Care — This condition is defined as usual care occurring within Community Based Outpatient Clinics (CBOCs), which typically does not involve substantial integration of mental health care and primary care.
  Other Names: Pre-Implementation
  Groups: Pre-Implementation Cohort
Other: Blended Telemedicine-Based Integrated Care — This condition involves exposure to a blended collaborative care model that includes care management for depression and alcohol disorders and "virtual co-location" of doctoral-level mental health providers with prompt access through tele-video or telephone communication.
  Other Names: Post-Implementation
  Groups: Post-Implementation Cohort

SUMMARY:
Integrating mental health treatments into the primary care delivered at Community Based Outpatient Clinics(CBOCs) that are geographically accessible to rural Veterans is a major priority for the Department of Veterans Affairs. However, there is no scientific evidence that integrating mental health and primary care is clinically effective at smaller CBOCs that have limited mental health staffing. The goal of this proposed project is to implement a "blended" combination of integrated care models that have been adapted for smaller CBOCs using telemedicine technologies, and evaluate the acceptability and effectiveness of the blended, telemedicine-based, integrated care model. If clinical outcomes are improved compared to usual care, findings will be used to justify and facilitate the implementation of this telemedicine-based integrated care model at smaller CBOCs in order to increase rural Veterans' access to effective mental health treatments.

DETAILED DESCRIPTION:
Background: Providing mental health care to rural Veterans in geographically accessible Community Based Outpatient Clinics (CBOCs) is a major priority of the Office of Rural Health. Likewise, integrating mental health into primary care is one of the highest priorities of the Office of Mental Health Services and the Office of Mental Health Operations. The Uniform Mental Health Services Handbook mandates the blending of the two predominant, evidence-based models of integrated care (the Care Management model and the Co-Located model) at VAMCs, very large CBOCs, and large CBOCs. Because there is no scientific evidence to support its implementation, the "Blended model" is not mandated at medium CBOCs or small CBOCs that serve rural Veterans. At most smaller CBOCs, on-site mid-level providers and/or off-site tele-psychiatrists and tele-psychologists deliver traditional referral-based specialty treatment (Referral model) rather than integrated care.

Objective: This project contributes to Specific Aim 3 (Test clinical interventions to improve quality and outcomes of mental health care at CBOCs) of the Little Rock CREATE application. The goal of this proposed Hybrid Type 2 pragmatic effectiveness-implementation trial is to generate the scientific evidence needed to justify the national dissemination of the Blended model adapted using telemedicine technologies to accommodate the clinical context of smaller CBOCs that lack on-site psychiatrists and PhD psychologists. The resulting Telemedicine Blended model will be compared to usual care (Referral model) in a pragmatic trial, where the intervention will be delivered via interactive video by centrally located clinical staff and fidelity will be monitored but not controlled. Specific Aim 1: Use an expert panel comprised of clinical providers and managers who are applying telemedicine to provide a Blended model for CBOCs lacking on-site PhD psychologists and psychiatrists to document the core components of a Telemedicine Blended model and using a PDSA process, implement this model in six CBOCs. Specific Aim 2: Conduct a Hybrid Type 2 pragmatic effectiveness-implementation trial of the adapted Telemedicine Blended model by assessing RE-AIM outcomes including: provider Reach into the patient population, Effectiveness at improving clinical outcomes, Adoption by providers and Implementation Fidelity.

Methods: In conjunction with national, regional and local partners, including providers and managers who have experience with the Telemedicine Blended model, the Blended model will be adapted for smaller CBOCs using telemedicine technologies and pilot tested to generate a standardized treatment protocol. We will use a stepped wedge design with randomization of sites to sequential implementation steps, and CBOC patients who screen positive for depression or alcohol disorders will be recruited and consented to participate in the Hybrid Type 2 pragmatic effectiveness-implementation trial. Data about Reach and Adoption will be obtained from the Corporate Data Warehouse. Data about Implementation Fidelity will be obtained from chart review. Data about clinical Effectiveness will be obtained from telephone survey.

Impact: If the Telemedicine Blended model improves clinical outcomes compared to usual care, results will be used to justify and facilitate the implementation of the Telemedicine Blended model at smaller CBOCs.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will enroll Veterans who screen positive on routinely administered VA mental health screens for depressive disorders, alcohol use disorders, and PTSD at the 6 study CBOCs.

Exclusion Criteria:

* Patients receiving specialty mental health treatment in the 6 months prior to recruitment and those who have a diagnosis of PTSD
* Those with a diagnosis of substance dependence
* Those with a psychotic disorder diagnosis:

  * schizophrenia
  * bipolar disorder
  * other psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be Veterans receiving care at 6 Community-Based Outpatient Clinics (primary care clinics) affiliated with the Central Arkansas Veterans Healthcare System or the Overton Brooks VA Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Owen, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR; JoAnn E. Kirchner, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Owen RR, Woodward EN, Drummond KL, Deen TL, Oliver KA, Petersen NJ, Meit SS, Fortney JC, Kirchner JE. Using implementation facilitation to implement primary care mental health integration via clinical video telehealth in rural clinics: protocol for a hybrid type 2 cluster randomized stepped-wedge design. Implement Sci. 2019 Mar 21;14(1):33. doi: 10.1186/s13012-019-0875-5. PMID 30898129
- [Result] Bauer MS, Miller C, Kim B, Lew R, Weaver K, Coldwell C, Henderson K, Holmes S, Seibert MN, Stolzmann K, Elwy AR, Kirchner J. Partnering with health system operations leadership to develop a controlled implementation trial. Implement Sci. 2016 Feb 24;11:22. doi: 10.1186/s13012-016-0385-7. PMID 26912342

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care (Pre-Implementation) Cohort: Eligible patients will be recruited and enrolled prior to implementation of the blended integrated care model in each study site. They will be exposed to care as usual in the CBOCs.
  Usual Care: This condition is defined as usual care occurring within Community Based Outpatient Clinics (CBOCs), which typically does not involve substantial integration of mental health care and primary care.
- Blended Telemedicine-Based Care (Post-Implementation) Cohort: Eligible patients will be recruited and enrolled following implementation of the blended integrated care model in each study site. These participants are thus exposed to the "intervention" model.
  Blended Telemedicine-Based Integrated Care: This condition involves exposure to a blended collaborative care model that includes care management for depression and alcohol disorders and "virtual co-location" of doctoral-level mental health providers with prompt access through tele-video or telephone communication.
Period: Overall Study
Arm/Group | Usual Care (Pre-Implementation) Cohort | Blended Telemedicine-Based Care (Post-Implementation) Cohort
Started | 279 | 39
Completed | 223 | 34
Not Completed | 56 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (Pre-Implementation) Cohort | Blended Telemedicine-Based Care (Post-Implementation) Cohort | Total
Number analyzed (Participants) | 279 | 39 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (14.8) | 48.9 (16.6) | 53.0 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 7 | 29
  Male | 257 | 32 | 289
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 272 | 38 | 310
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 93 | 7 | 100
  White | 165 | 32 | 197
  More than one race | 17 | 0 | 17
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 279 | 39 | 318
VR-12 MCS [Mean (Standard Deviation); unit: units on a scale] — The Veterans RAND 12-Item Health Survey (VR-12) Mental Component Summary (MCS) is a normed scale, presented as a T-score that is standardized to the US population. The population mean MCS score is 50 and standard deviation is 10, with scores ranging from 0-100. A higher score represents better mental health-related quality of life. A score of 30 signifies that the MCS score is two standard deviations below the population mean. The VR-12 was developed from the Veterans RAND 36-Item Health Survey (VR-36), which was developed from the Medical Outcomes Study RAND SF-36(TM) Version 1.0.
  units on a scale | 39.7 (13.5) | 38.2 (13.7) | 39.5 (13.5)
VR-12 PCS [Mean (Standard Deviation); unit: units on a scale] — The Veterans RAND 12-Item Health Survey (VR-12), Physical Component Summary (PCS) is a normed scale, presented as a T-score that is standardized to the US population. The population mean PCS score is 50 and standard deviation is 10, with scores ranging from 0-100. A higher score represents better health-related quality of life. A score of 30 indicates that the PCS score is two standard deviations below the population mean. The VR-12 was developed from the Veterans RAND 36-Item Health Survey (VR-36), which was developed from the Medical Outcomes Study RAND SF-36(TM) Version 1.0.
  units on a scale | 32.7 (13.6) | 36.8 (13.6) | 33.2 (13.6)
Marital Status [Count of Participants; unit: Participants] — Marital status - categorized dichotomously as married or living with someone; or all other statuses.
  Participants | 164 | 23 | 187
Education [Count of Participants; unit: Participants] — Education - trichotomous categorical variable: (1) high school or less; (2) some college; (3) college degree or more.
  Participants
    High School or Less | 107 | 8 | 115
    Some College | 118 | 13 | 131
    College Degree or More | 54 | 18 | 72
Employment [Count of Participants; unit: Participants] — Employment status, categorized as (1) full-time or part-time; (2) retired; (3) other.
  Participants
    Full-Time or Part-Time | 98 | 21 | 119
    Retired | 73 | 6 | 79
    Other | 108 | 12 | 120
Non-VA Health Insurance Status [Count of Participants; unit: Participants] — Any health insurance reported, not including VA eligibility/enrollment.
  Participants | 163 | 21 | 184
Clinical Depression Screen Positive [Count of Participants; unit: Participants] — Depression screening test, administered as part of routine clinical care, is positive. Typical depression screener is PHQ-2.
  Participants | 116 | 17 | 133
Clinical Alcohol Screening Test - Positive [Count of Participants; unit: Participants] — Number of participants with a positive alcohol screening test (typically AUDIT-C) administered as part of routine clinical care.
  Participants | 106 | 22 | 128
Clinical PTSD Screening - Positive [Count of Participants; unit: Participants] | 105 | 1 | 106
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire-9 (PHQ-9) total score at baseline. The possible range of scores is 0-27, with higher scores indicating more severe depressive symptoms.
  units on a scale | 11.2 (6.3) | 11.3 (6.3) | 11.2 (6.3)
AUDIT-C Total Score [Mean (Standard Deviation); unit: units on a scale] — Alcohol Use Disorders Identification Test (AUDIT-C) Total Score. The possible range of scores is 0-12, with higher scores indicating greater alcohol use.
  units on a scale | 3.6 (3.5) | 4.6 (2.9) | 3.8 (3.4)
PCL-5 [Mean (Standard Deviation); unit: units on a scale] — PTSD Checklist for DSM-5 Total Score. Possible scores range from 0-80, with higher scores indicating greater symptom severity.
  units on a scale | 30.4 (17.6) | 29.2 (17.4) | 30.3 (17.6)
Hoge Barriers Assessment [Mean (Standard Deviation); unit: units on a scale] — Hoge Barriers Assessment Total Score. The possible range of scores is 14-70, with higher scores indicating greater barriers.
  units on a scale | 33.9 (8.8) | 33.1 (9.9) | 33.8 (8.9)
Readiness Ruler [Median (Inter-Quartile Range); unit: units on a scale] — Readiness Ruler: Assessment of Motivation for Treatment for Any Mental Health Concern. Readiness 1: "How important...to receive treatment..."; Readiness 2: "How confident...that you would get treatment"; Readiness 3: "How ready are you to receive treatment..." Each question is rated on a scale of 0-10, with higher scores indicating greater importance, confidence, and readiness, respectively. Population: There were missing data for Readiness 2 and Readiness 3 measures for a few participants.
  units on a scale
    Readiness 1 | 6.0 [2.0 to 8.0] | 7.0 [5.0 to 9.0] | 6.0 [2.0 to 8.0]
    Readiness 2: number analyzed (Participants) | 273 | 38 | 311
    Readiness 2 | 8.0 [5.0 to 10.0] | 8.0 [6.0 to 10.0] | 8.0 [5.0 to 10.0]
    Readiness 3: number analyzed (Participants) | 276 | 39 | 315
    Readiness 3 | 7.0 [4.0 to 10.0] | 8.0 [5.0 to 10.0] | 7.0 [4.0 to 10.0]
Pain Scale [Mean (Standard Deviation); unit: units on a scale] — Single item participant rating of the average overall level of pain for the past week rated on a continuous scale from 0 to 10, with higher ratings indicating more severe pain.
  units on a scale | 5.1 (2.7) | 4.8 (2.9) | 5.1 (2.7)
Jenkins Sleep Scale [Median (Inter-Quartile Range); unit: units on a scale] — Jenkins Sleep Scale, a four-item measure that assesses trouble falling and staying asleep. Possible scores range from 0-20, with higher ratings indicating more substantial sleep problems. Population: Missing data for 8 participants in the pre-implementation participant group.
  units on a scale
    number analyzed (Participants) | 271 | 39 | 310
    (all) | 14.0 [8.0 to 18.0] | 16.0 [8.0 to 18.0] | 14.0 [8.0 to 18.0]
GAD-7 [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder Scale, a 7 item inventory that yields a continuous and dichotomous assessment of generalized anxiety disorder. Possible scores range from 0-21, with scores of 10 or greater indicating a positive screen for generalized anxiety disorder.
  units on a scale | 9.1 (6.0) | 10.4 (6.1) | 9.3 (6.0)
Severity Measure for Panic - Adult [Mean (Standard Deviation); unit: units on a scale] — American Psychiatric Association DSM-5 Severity Measure for Panic - Adult - 10 item inventory that yields a continuous and dichotomous assessment of panic disorder. Possible scores range from 0-28, with higher scores indicating more severe symptoms. Population: Total score presented here only applies to participants who reported ever having a panic attack.
  units on a scale
    number analyzed (Participants) | 142 | 22 | 164
    (all) | 12.1 (8.6) | 10.6 (8.6) | 11.9 (8.6)
BRFSS Tobacco Use [Count of Participants; unit: Participants] — The Behavioral Risk Factor Surveillance System (BRFSS) Tobacco Use measure was administered. It has 5 items to assess current tobacco use, with a dichotomous variable being created to indicate any tobacco use. Population: This item was assessed for participants who answered the first question, "Have you smoked at least 100 cigarettes in your entire life?" in the affirmative.
  Participants
    number analyzed (Participants) | 197 | 24 | 221
    (all) | 109 | 10 | 119
CSQ-8 [Median (Inter-Quartile Range); unit: units on a scale] — The Client Satisfaction Questionnaire-8 (CSQ-8) consists of 8 items to assess participant satisfaction with mental health services. Possible scores range from 8-32, with higher scores indicating greater client satisfaction. Population: One participant in the pre-implementation participant group had missing data on this scale.
  units on a scale
    number analyzed (Participants) | 278 | 39 | 317
    (all) | 27.0 [23.0 to 31.0] | 28.0 [25.0 to 30.0] | 27.0 [23.0 to 30.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in VR-12 Mental Component Summary Scores
Description: Change in overall mental health functioning from study enrollment (after screening positive for depressive disorder or alcohol use disorder) to six-month follow-up on the Mental Component Summary scale of the Veterans Rand 12-item Health Survey. Measure Description: The Veterans RAND 12-Item Health Survey (VR-12) Mental Component Summary (MCS) is a normed scale, presented as a T-score that is standardized to the US population. The population mean MCS score is 50 and standard deviation is 10, with scores ranging from 0-100. A higher (positive) change score represents greater improvement in mental health-related quality of life from study enrollment to follow-up. The VR-12 was developed from the Veterans RAND 36-Item Health Survey (VR-36), which was developed from the Medical Outcomes Study RAND SF-36(TM) Version 1.0.
Time Frame: Six months
Population: The number of participants analyzed for each cohort is somewhat less than the number of total participants in each group (1) because of loss to follow-up and (2) because participants who only screened positive for PTSD were not included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (Pre-Implementation) Cohort | Blended Telemedicine-Based Care (Post-Implementation) Cohort
Number analyzed (Participants) | 172 | 33
score on a scale | 2.9 (11.8) | 5.1 (9.6)

2. Secondary Outcome: Change in PHQ-9 Scores
Description: Change in depressive symptoms as measured by Patient Health Questionnaire (PHQ-9) from study enrollment to six-month follow-up, for patients screening positive for depressive disorders at baseline. The possible range of scores on the PHQ-9 is 0-27, with higher scores indicating more severe depressive symptoms. A negative change score represents improvement in depressive symptoms.
Time Frame: Six months
Population: The numbers of participants analyzed in each cohort for this measure is less than the total number of participants (1) because this analysis only included participants who had screened positive for depression and (2) because of loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (Pre-Implementation) Cohort | Blended Telemedicine-Based Care (Post-Implementation) Cohort
Number analyzed (Participants) | 116 | 17
score on a scale | -2.3 (6.0) | -3.2 (3.8)

3. Secondary Outcome: Change in AUDIT-C Scores
Description: Change in alcohol use symptoms from study enrollment to six-month follow-up, for patients screening positive for alcohol use disorders at baseline. The analysis used the Alcohol Use Disorders Identification Test (AUDIT-C) Total Score. The possible range of scores is 0-12, with higher scores indicating greater alcohol use.
Time Frame: Baseline, Six months
Population: Participants are included in this analysis if they screened positive for alcohol use disorder (clinical screen) before enrollment. The number of participants analyzed is lower than the total enrolled in the study because many participants did not screen positive for alcohol use disorder. At 6-month follow-up assessment, some participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
Number analyzed (Participants) | 106 | 22
units on a scale
  Baseline assessment | 6.8 (2.8) | 6.5 (1.7)
  6-month follow-up assessment: number analyzed (Participants) | 88 | 21
  6-month follow-up assessment | 6.4 (2.7) | 6.1 (2.0)

4. Other Pre Specified Outcome: Adoption of Intervention by Primary Care Providers
Description: Proportion of primary care providers with at least one patient with a Primary Care-Mental Health Integration encounter following implementation of the blended, integrated care model. The time frame is variable due to the stepped wedge design.
Time Frame: 12-24 months
Reporting Status: Not Posted, anticipated posting 2025-02

5. Other Pre Specified Outcome: Reach of Intervention
Description: Proportion of patients having any mental health encounter in the six month follow-up period.
Time Frame: Six months
Reporting Status: Not Posted, anticipated posting 2025-04

ADVERSE EVENTS:
Time Frame: Each participant was followed for 6 months after enrollment.
Description: We are using the clinicaltrials.gov definitions.
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
All-Cause Mortality (participants affected / at risk) | 1/279 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/279 | 0/39
Other Adverse Events (participants affected / at risk) | 0/279 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT02713217/Prot_SAP_000.pdf